CLINICAL TRIAL: NCT04854187
Title: The Effect of Personal Protective Aids on Hypertension and Diabetes in People Exposed to High Levels of Air Pollution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Indian Institute of Technology Kanpur (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IITK/IEC/2020-21/II/31
Record Dates: First submitted 2021-03-30; First posted 2021-04-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Pollution; Exposure; HTN; Diabetes Mellitus
Keywords: Air pollution; HTN; DM; N95 mask; Indoor air purifier
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Prospective, randomized cross over study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Arm - Indoor air purifier and N95 mask (Active Comparator): Intervention arm will be for 4 weeks. Blood pressure and/or blood glucose will be recorded on day 0; end of week 2 and end of the intervention. Participants in the intervention group will be asked to use an indoor air purifier (Atlanta Healthcare 7-Stage 43-Watt Air Purifier) daily for 4 weeks between the hours of ¬8 PM and 8 AM. The purifier will be placed in their bedroom or in the room where participants sleep at night. When the participants are outdoors (commuting, working outdoors, running errands, etc.), they will be asked to use a N95 mask (PureMe Reusable N95 Anti-Pollution Mask). It is a reusable mask which can be washed by the participants. Every 2 weeks, the filter of the mask will be replaced, and the filter of the indoor purifier will be washed.
  Interventions: Device: N95 Mask/Indoor air purifier: Including sham
- Washout period - No intervention (No Intervention): At the end of either control or intervention arm, participants will have a washout period of 2 weeks, after which participants will be crossed over to the other group for the subsequent 4 weeks. For example, after Participant AB is in intervention arm for 4 weeks, he/she will then have a wash out period of 2 weeks in which they will return to their usual state of living. At the end of the washout period, the participant AB will be put in the control arm for 4 weeks.
- Controlled Arm - Indoor air purifier and N95 mask with sham filter (Sham Comparator): Control arm will be for 4 weeks. Blood pressure, blood glucose and indoor air pollution level will be recorded similarly as in the intervention group on day 0, end of week 2 and week 4. The participant will be provided an air purifier and a N-95 mask (of the same manufacturer), with the filter removed. At the end of two weeks, the health worker will make dummy adjustments to the mask and indoor air purifier, to maintain blinding of the participant.
  Interventions: Device: N95 Mask/Indoor air purifier: Including sham

INTERVENTIONS:
Device: N95 Mask/Indoor air purifier: Including sham — Participants will be using indoor air purifier and N95 mask (control arm with sham filters). The effect will be studied on blood pressure and blood glucose levels.
  Arms: Controlled Arm - Indoor air purifier and N95 mask with sham filter; Intervention Arm - Indoor air purifier and N95 mask

SUMMARY:
This is a randomized controlled trial to evaluate personal protective aids (air purifier and N95) as a therapeutic measure in people with hypertension and diabetes exposed to high levels of PM2.5 in India.

DETAILED DESCRIPTION:
Air pollution is the largest environmental cause of disease and premature death in the world today, disproportionally affecting low- and middle-income countries (LMICs) such as India. Numerous studies have shown that exposure to particulate matter <2.5 µm (PM2.5) can contribute to cardiovascular disease and mortality, which is partially attributable to the development of cardiometabolic conditions such as hypertension and diabetes. We hypothesize that the use of personal protective aids (home air-purifier and N-95 mask) can decrease systolic blood pressure (SBP) in people with hypertension and decrease fasting blood glucose (FBG) in those with diabetes.

This is a prospective randomized cross-over study in Dalkhola, India- an area of high ambient PM2.5 levels. Participants between 18 and 70 years of age with hypertension (n=130) and diabetes (n=33) will be invited to participate in the study. They will be randomized to either an intervention or control arm for 4 weeks, after which they will cross over to the other arm following a 2-week washout period. The intervention period will consist of using an indoor air-purifier at night and an N-95 mask when outdoors. Control period will involve using an identical air purifier and facemask, with the filter removed (sham filtration). Participants and outcome assessors will be blinded.

The primary outcome of the study is the absolute reduction in SBP among people with hypertension and absolute reduction in FBG among people with diabetes.

This is the first randomized controlled trial to evaluate personal protective aids as a therapeutic measure in people with hypertension and diabetes exposed to high levels of PM2.5. Given the high burden of air pollution in LMICs, there is an urgent need for adaptation measures targeting people at high risk for mortality from this exposure. The results of our study will demonstrate if personal protective aids can be a viable adaptation measure for people living with hypertension and diabetes in areas with a high burden of air pollution.

ELIGIBILITY:
Inclusion Criteria:

Hypertension arm

1. Individuals age 18-70 years old with systolic blood pressure between 130-160 mmHg, regardless of medication use
2. Stable hypertension for the past 3 months with no medication changes
3. No planned medication changes for the duration of the study
4. Exposure to outdoor air pollution above a certain threshold (pollution levels will be measured using AirVeda devices)
5. Individuals who sleep in a closed space (such as a bedroom) for minimum of 6 hours/daily.
6. Use of gas (LPG)/electricity for cooking purposes

Diabetes arm

1. Individuals age 18-70 years old with fasting blood glucose between 126-180 mg/dL, regardless of medication use
2. Stable diabetes for the past 3 months with no medication changes
3. No planned medication changes for the duration of the study
4. Exposure to outdoor air pollution above a certain threshold (pollution levels will be measured using AirVeda devices)
5. Individuals who sleep in a closed space (such as a bedroom) for minimum of 6 hours/daily.
6. Use of gas (LPG)/electricity for cooking purposes

Exclusion Criteria:

1. Unwilling to participate
2. Unstable blood pressure and/or blood glucose level requiring frequent medication changes
3. Individual suffering from a physical or mental illness that precludes active study participation
4. Current smoker
5. Planned vacation/absence from the study site
6. Patients with life expectancy < 12 months
7. Pregnant patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Absolute change in systolic blood pressure for people with hypertension using air purifier and facemask | 4 weeks
  We will monitor blood pressure at week 0,2,4 of both intervention and control period. Outcome would be measured as difference in the mean systolic blood pressure between both arms.
Absolute change in fasting blood glucose for people with diabetes using air purifier and facemask | 4 weeks
  We will monitor fasting blood glucose at week 0,2,4 of both intervention and control period. Outcome would be measured as difference in the mean systolic blood pressure between both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Dweep Barbhaya, MD, Principal Investigator — Medstar Health Research Institute; Aditya Khetan, MD, Principal Investigator — Hamilton Health Sciences, McMaster University, Hamilton, Canada
Locations (1):
- Sehat Charitable trust, Dalkhola, West Bengal, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barbhaya D, Tran J, Khetan A, Hejjaji V, Jain S, Chan C, Goel A. Rationale and Design of a Study to Test the Effect of Personal Protective Aids on Hypertension and Diabetes in People Living With High Levels of Air Pollution-Study Protocol. Heart Lung Circ. 2023 Jan;32(1):124-130. doi: 10.1016/j.hlc.2022.11.001. Epub 2022 Dec 15. PMID 36528547

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT04854187/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT04854187/ICF_001.pdf